CLINICAL TRIAL: NCT01322867
Title: A Phase IV, Open Label, Randomized, Two-way Crossover, Single Dose Study to Determine Relative Bioavailability of Alprazolam 0,75mg/ml (laboratórios Pfizer Ltda) in the Oral Solution-drops Form, Versus Frontal® 0,25mg (laboratórios Pfizer Ltda), in the Tablets Form, Under Fasted Conditions in Healthy Volunteers.
Brief Title: A Bioequivalence Study Of A New Alprazolam Dropped Formulation Versus Alprazolam Tablets
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: A6131023
Record Dates: First submitted 2011-03-23; First posted 2011-03-25 (Estimated); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Healthy
Keywords: bioequivalence study; alprazolam; frontal
MeSH Terms: interventions — Alprazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Reference Drug (Active Comparator)
  Interventions: Drug: alprazolam tablet
- Test Drug (Active Comparator)
  Interventions: Drug: alprazolam oral solution

INTERVENTIONS:
Drug: alprazolam tablet — 0,25 mg oral tablets given once
  Arms: Reference Drug
Drug: alprazolam oral solution — 0,75 mg/ml Oral Solution (Drops) given once
  Arms: Test Drug

SUMMARY:
A Phase IV, Open Label, Randomized, Two-way Crossover, Single Dose Study to Determine Relative Bioavailability of Alprazolam 0,75mg/ml (laboratórios Pfizer Ltda) in the Oral Solution-drops Form, Versus Frontal® 0,25mg (laboratórios Pfizer Ltda), in the Tablets Form, Under Fasted Conditions in Healthy Volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects between the ages of 18 and 55 years, inclusive (Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12-lead ECG and clinical laboratory tests)
* The BMI - Body Mass Index of the volunteers should be within the range of 18,5 to 24,9 (Dietary Guidelines for Americans) and it may vary up to 15% due to the upper limit (18,5 to 28,63) and total body weight >50kg
* An informed consent document signed and dated by the subject or a legally acceptable representative. If the subject and/or legally acceptable representative cannot read, then the informed consent document may be signed by an impartial witness
* Subjects who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures

Exclusion Criteria:

* Any condition possibly affecting drug absorption (eg, gastrectomy)
* A history of suicidal thoughts, behavior or suicide attempts
* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing)
* Known hypersensitivity to alprazolam or any components of the product
* History of sensitivity to heparin or heparin-induced thrombocytopenia
* A positive bHCG exam for women
* Subjects with myasthenia gravis or acute narrow angle glaucoma

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2011-05; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) of Test Drug and Reference Drug | Up to 72h
Area under the plasma concentration versus time curve from time zero to the last measurable concentration of Test Drug and Reference Drug (AUC(0-tlast)) | Up to 72h

SECONDARY OUTCOMES:
Area under the plasma concentration versus time curve from time zero to infinity of Test Drug and Reference Drug (AUC(0-inf)) | Up to 72h
Time to peak concentration of Test Drug and Reference Drug (Tmax) | Up to 72h
Half-life of Test Drug and Reference Drug (T1/2) | Up to 72h
Elimination rate constant (K el) | Up to 72h
Area under the curve from the time of dosing (AUC t/inf) extrapolated to infinity | Up to 72h

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- ICF - Instituto de Ciencias Farmaceuticas, Aparecida de Goiânia, Goiás, Brazil

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6131023&StudyName=A%20Bioequivalence%20Study%20Of%20A%20New%20Alprazolam%20Dropped%20Formulation%20Versus%20Alprazolam%20Tablets